CLINICAL TRIAL: NCT05170035
Title: Autologous Patch Healing vs. Secondary Intention Healing After Mohs Micrographic Surgery - A Randomized Controlled Trial
Brief Title: Autologous Patch Healing vs. Secondary Intention Healing After Mohs Micrographic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Benzon Foundation (Unknown)
Responsible Party: Principal Investigator, Katrine Elisabeth Karmisholt, MD, Chief Consultant, Ass.Prof., PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Autologous Patch-project
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Skin Cancer; Basal Cell Carcinoma
Keywords: Skin Cancer; Basal Cell Carcinoma; Mohs micrographic surgery; MMS; Autologous patch; Secondary intention healing
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Blinded photo assesment of wound healing by two independent trained clinical doctors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMS + Autologous patch (Experimental): Mohs micrographic surgery + Autologus patch formed from 18 ml venous blood sample collected from the patient + polymycin-terramycin B ointment and a Jelonet applied on top of the patch.
  Interventions: Procedure: MMS + Autologous patch
- MMS + Secondary intention healing (Active Comparator): Mohs micropgraphic surgery + Polymycin-terramycin B ointment + dry wound dressing
  Interventions: Procedure: MMS and secondary intention healing

INTERVENTIONS:
Procedure: MMS + Autologous patch — A patch of consisting of platelets, leucocytes and fibrin, formed by the patients own blood sample.
  Arms: MMS + Autologous patch
Procedure: MMS and secondary intention healing — Mohs micrographic surgery (standard of care) (wounds will heal by secondary intention healing)
  Arms: MMS + Secondary intention healing

SUMMARY:
The primary objects of this study is to explore the potential effect of the autologous patch to optimize wound healing after skin cancer surgery with Mohs micrographic surgery (MMS) in the face in a randomized controlled trial comparing autologous patch healing versus secondary intention healing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing MMS for biopsy verified primary nodular basal cell carcinoma in the face, head and neck area on a location suitable for secondary intention healing and thus may also be suitable for autologous patch healing
2. Presenting relevant medical record report at study initiation
3. Written informed consent obtained from subject
4. Understanding of investigation procedures and willingness to abide to all procedures during the course of the investigation.

Exclusion Criteria:

1. A subjects with major systemic disease not yet stabilized
2. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
3. Pregnant or breast feeding
4. Unable to follow the outlined study protocol
5. Participation in other studies at the same time that may affect the wound healing.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Blinded assesment of wound healing at day 18-20. | Day 18-20
  Two indenpendent trained clinical doctors will evaluate clinical photos. Wounds will be evaluated fully epithelialized yes/no.

SECONDARY OUTCOMES:
Blinded assesment of wound healing at day 11-13 | day 11-13
  Clinical photos from day 11-13 will be evaluated. Wounds will be evaluated 50% fully epithelialized yes/no.
TEWL measurement | day 11-13 and day 18-20
  Trans epidermal water loss (TEWL) will be meassured at day 11-13 and day 18-20. The TEWL will be meassured on the wound healing site and the contralateral site of the patient's face as a control.
Scar evaluation using the patient-observer-scar-assesment-scale (POSAS) at 6 months follow-up. | 6 months
  The POSAS observer scores scar components with regards to: Vascularity, pigmentation, thickness, surface area, relief and pliability. The collected sum of scores will range from minimum 6 points to maximum 60 points.
Difference in microbiology between intervention wounds and control wounds. | day 1 and day 11-13
  Swab test for microbiome analysis will be conducted at day 1 and day 11-13.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark